CLINICAL TRIAL: NCT07403331
Title: Optimizing Treatment for Chronic Neuropathic Pain: A Replicated Single Case Experimental Design Evaluating a Treatment Bundle Consisting of Multidisciplinary Rehabilitation and Spinal Cord Stimulation (SCS-R)
Brief Title: Severe Chronic Neuropathic Pain: A Treatment Bundle, Using Spinal Cord Stimulation and Multidisciplinary Treatment, to Reduce Pain and Improve Physical Function.
Acronym: SCS-R
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars-Petter Granan, Head of Department, Department for pain management and research. Ph.D., Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 942321
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neuropathic Pain; Multidisciplinary Approach; Rehabilitation Exercise; Acceptance & Commitment Therapy; Spinal Cord Stimulation (SCS)
MeSH Terms: conditions — Neuralgia | interventions — Spinal Cord Stimulation; Rehabilitation; Acceptance and Commitment Therapy; Cognitive Behavioral Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The study examines a treatment bundle consisting of spinal cord stimulation plus multidisciplinary rehabilitation. We use a single-case experimental design (SCED) which is based on N-of-1 trials: each participant acts as their own control. A long baseline period with many measurement points establishes a stable baseline. The same is done during the intervention, and at 6-month follow-up.
  We repeat this structure across10 participants, and combine individual effects to estimate a pooled treatment effect while keeping within-person precision.
  Randomization is used only for baseline length (5, 6, or 7 weeks), creating a multiple-baseline design to strengthen causal inference.
  There is no separate control group; each participant's baseline serves as the comparison.
  SCEDs suit this study because the intervention is complex, and because chronic pain also is complex.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment bundle (Experimental): Treatment bundle consisting of spinal cord stimulation plus multidisciplinary rehabilitation
  Interventions: Other: Treatment bundle

INTERVENTIONS:
Other: Treatment bundle — The intervention is a treatment bundle consisting of spinal cord stimulation plus multidisciplinary rehabilitation. The multidisciplinary rehabilitation consists of excercise therapy, cognitive therapy and individualized programming of the SCS device.
  Other Names: Spinal cord stimulation; Rehabilitation; Excercise therapy; Acceptance and commitment therapy; Cognitive therapy; Physiotherapy

SUMMARY:
People with nerve damage can develop nerve pain. The pain can sometimes be severe and unpredictable, causing odd or alarming sensations - for example, lightning-like or electric shock feelings in the area served by the damaged nerve.

We will examine a treatment for nerve pain in the legs caused by nerve damage, which can occur after a herniated disc or a bone fracture, with or without surgery.

Previous research suggests that spinal cord stimulation can relieve nerve pain in the legs after surgery or injury, but its effectiveness is still debated. Other studies show that multidisciplinary treatment helps people with long-term pain to improve their quality of life and to better cope in life. National and international guidelines recommend this kind of multidisciplinary care for long-term pain.

No one has yet published research on spinal cord stimulation combined with multidisciplinary treatment as a bundle intervention. We therefore want to find out whether this combined approach can reduce nerve pain in the legs and improve physical functioning.

ELIGIBILITY:
Inclusion criteria:

* Peripheral neuropathic pain in one or both legs for >6 months due to:

  * (1) Post Spinal Pain Syndrome (type 1 or 2).
  * (2) Localized nerve damage.
* The area of the neuropathic pain in the leg(s) must be the dominant pain component.
* Age ranges from 18-60 years.
* Previous standard conservative (or surgical) treatment attempted.
* Opioid use within permissible limits at implantation time (daily opioid dose <50 mg OMEQ).
* Willingness to actively participate in the treatment bundle.
* Living within reasonable travelling distance from Oslo.
* Proficiency in understanding oral and written Norwegian, essential to benefit from the program that relies on mutual comprehension, nuanced conversation, and emotional expression, which are language-dependent.
* Cognitive capacity to provide informed consent.
* Ability to master the technical aspects of the SCS system (switching programs on the remote control).

Exclusion criteria:

* Currently undergoing the claims process for health benefits (e.g., disability pensions from NAV (Norwegian Labour and Welfare Administration).
* Presenting a psychological or psychiatric disorder that may impact treatment efficacy.
* Chronic generalized pain conditions.
* Other pain conditions in the affected area, such as osteoarthritis.
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity in leg(s) | 3 times per week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  Assessed using an 11-point Numeric Rating Scale (NRS 0-10), where 0 = "no pain" and 10 = "worst imaginable pain." Higher scores indicate more severe pain.
Physical function | 3 times per week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  PROMIS-29 Physical Function domain, reported as a T-score (higher scores indicate better function).

SECONDARY OUTCOMES:
Pain intensity in the lower back | 3 times per week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  Assessed using an 11-point Numeric Rating Scale (NRS; 0-10), where 0 = "no pain" and 10 = "worst imaginable pain." Higher scores indicate greater pain intensity.
Physical function | Once pre-implantation, at end of intervention (approximately 12 weeks post-implantation), and once during follow-up period at 6 months post-implantation.
  6-minute walk test (6MWT; total distance walked in meters; higher values indicate better physical function).
Physical function | Once pre-implantation, at end of intervention (approximately 12 weeks post-implantation), and once during follow-up period at 6 months post-implantation.
  30-second sit-to-stand test (30sSTS; number of stands completed; higher values indicate better function).
Physical function | Once pre-implantation, at end of intervention (approximately 12 weeks post-implantation), and once during follow-up period at 6 months post-implantation.
  Stair test (ST; time to climb 18 stairs 3 times; lower times indicate better function).
Health-related quality of life (index) | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  EQ-5D-5L index score (range 0-1; higher scores indicate better health-related quality of life).
Health-related quality of life (VAS) | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  EQ-5D Visual Analogue Scale (EQ-5D VAS; 0-100; higher scores indicate better health-related quality of life).
Depression symptoms | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  PROMIS Depression scale (T-score; mean 50, SD 10 in U.S. population; higher scores indicate greater symptom severity).
Social participation | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  PROMIS Ability to Participate in Social Roles and Activities short form, reported as a T-score (higher scores indicate better function).
Fatigue | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  PROMIS Fatigue scale, reported as a T-score (higher scores indicate greater fatigue severity).
Pain interference | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  PROMIS Pain Interference scale, reported as a T-score (higher scores indicate greater pain interference).
Sleep disturbance | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  PROMIS Sleep Disturbance scale, reported as a T-score (higher scores indicate greater sleep disturbance).
Opioid and Analgesic Use | Once pre-implantation, at end of intervention (approximately 12 weeks post-implantation), and once during follow-up period at 6 months post-implantation.
  Total opioid consumption quantified as milligrams of oral morphine equivalents (OMEQ) per day; non-opioid analgesics quantified in milligrams per day per medication.
Return to work | Once pre-implantation, at end of intervention (approximately 12 weeks post-implantation), and once during follow-up period at 6 months post-implantation.
  Return to work status, quantified as hours worked per week (higher values indicate greater work participation).
Fear of movement | Once pre-implantation, at end of intervention (approximately 12 weeks post-implantation), and once during follow-up period at 6 months post-implantation.
  Tampa Scale of Kinesiophobia (TSK; total score 13-52; higher scores indicate greater kinesiophobia).
Patient-specific functioning | Once a week during (A) baseline period (randomized length: 5, 6, or 7 weeks), (B) intervention period (12 weeks), and (C) follow-up period (5 weeks) at 6 months post-implantation.
  Patient-Specific Functional Scale (PSFS), up to five activities selected in cooperation with personnel, rated 0-10 (higher scores indicate better function; average score reported).
Patient satisfaction | Measured at end of intervention (approximately 12 weeks post-implantation) and 26-week follow-up (6 months post-implantation).
  Patient Global Impression of Change (PGIC), 7-point Likert scale (1 = "very much worse" to 7 = "very much improved").

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Petter Granan, Ph.D, Principal Investigator — Department of pain management and research, Oslo university hospital
Locations (1):
- Department of pain management and research, Oslo university hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all collected variables, generated during the study and fully documented in an accompanying data dictionary (detailing variable names, codes, values, units, and derivations), will be made available upon reasonable request from qualified researchers after publication Access will be restricted to qualified researchers who submit an application and obtain approval from the relevant ethics committee and data protection authority.
  Direct and indirect identifiers-including names, exact dates, and other re-identification risks-will be systematically removed or transformed (such as index-adjusting dates to retain intervals while preventing linkage), ensuring the dataset supports robust secondary analyses while upholding participant privacy.
  The study protocol is planned to be published.